CLINICAL TRIAL: NCT05707884
Title: Prospective Evaluation of Volatile Sedation Management in Critical Care After Free Flap Surgery
Brief Title: Volatiles in Critical Care After Free Flap Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Armin N. Flinspach, Principal Investigator, Goethe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-1040
Record Dates: First submitted 2022-12-27; First posted 2023-02-01 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2023-10

CONDITIONS: Sedation Set-up Time; Additional Time Required for Volatile Sedation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- volatile sedation (Active Comparator): Patients receive volatile sedation for the intended 72 hours of deep sedation after complex free flap surgery.
  Interventions: Other: critical care management
- intravenous sedation (No Intervention): Patients receive intravenous sedation (e.g. propofol) for the intended 72 hours of deep sedation after complex free flap surgery.

INTERVENTIONS:
Other: critical care management — The different sedation methods result in considerable differences in terms of set-up costs and the management of the patient, which will be examined in a direct comparison.
  Arms: volatile sedation

SUMMARY:
Patients undergoing complex free flap surgery are randomised to volatile or intravenous sedation in terms of subsequent intensive care sedation, based on the in-hospital standard of care. For study purposes, differences in management (set-up times, change of filters, etc.) will be investigated in relation to accelerated awakening and possibly improved neurocognition after the end of sedation.

ELIGIBILITY:
Inclusion Criteria:

* Free flap surgery
* Patient capable of giving informed written consent

Exclusion Criteria:

* Intolerance to volatile anaesthetics (e.g. malignant hyperthermia).
* Severe obstructive pulmonary disease
* Pre-existing severe neurocognitive disorder
* Age <18 years (minors)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Material consumption | Inventory of the required materials until the end of sedation (90 hours)
  Required equipment and disposable materials related to the treatment interval as well as their monetary value in euros or US dollars.
Working time expenditure | Inventory of the required time until the end of sedation (90 hours)
  Time spent by nurses or physicians on the specific sedation procedure, as well as the corresponding financial value based on nationally applicable collective wage agreements in euros or US dollars.

SECONDARY OUTCOMES:
Delir | Within the intensive care stay (5 days)
  Occurrence of delirium in the intensive care setting
Time to awake | Within the intensive care stay (5 days)
  Time required beyond the intended 72 hours of sedation for the patient to awaken

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No